CLINICAL TRIAL: NCT04998682
Title: TAD: Prospective Evaluation of Targeted Axillary Dissection After Neoadjuvant Systemic Therapy in Patients With Breast Cancer With Advanced Nodal Disease at Diagnosis
Brief Title: Prospective Evaluation of Targeted Axillary Dissection (TAD)
Acronym: TAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Susan Kesmodel, MD, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201540; NCI-2021-11060 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2021-08-07; First posted 2021-08-10 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Targeted Axillary Dissection; Advanced Nodal Disease; Axillary Lymph Node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Targeted Axillary Dissection (TAD) (Experimental): During standard of care (SoC) surgery to remove breast cancer, study participants will undergo a sampling of lymph nodes in the axilla first and then complete removal of axillary lymph nodes under the arm.
  Interventions: Procedure: Axillary Dissection

INTERVENTIONS:
Procedure: Axillary Dissection — A surgical procedure that opens the armpit (axilla) to identify, examine, or remove lymph nodes. Axillary dissection will be performed during SoC breast cancer surgery.

SUMMARY:
The purpose of this research is to evaluate how to manage the axillary lymph nodes in patients with breast cancer. The investigators will determine if a sampling of the lymph nodes under the arm will give the information necessary to determine if fewer lymph nodes can be removed.

ELIGIBILITY:
Inclusion Criteria:

* Women or men greater than or equal to 18 years.
* Histologically confirmed invasive adenocarcinoma of the breast.
* Clinical T0-4 N2-3 M0 at diagnosis (American Joint Committee on Cancer, 7th Edition)

  * Assessment for cN2 disease will be performed by clinical exam and imaging. Patients should have pathologic level 1 and/or 2 axillary lymph nodes which are fixed/matted on physical exam.
  * Cross-sectional imaging will be used to identify advanced nodal disease involving the axilla, infraclavicular, supraclavicular, and internal mammary regions, cN3 disease.
* Patients must have biopsy proven involvement of the axillary lymph nodes.
* Receipt of standard multiagent chemotherapy +/- targeted therapy based on tumor subtype.
* Candidate for surgical management of breast cancer.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions or hypersensitivity to radioactive lymph node mapping agents or blue dye.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
False Negative Rate | Up to 2 weeks
  The false negative rate of targeted axillary dissection after neoadjuvant systemic therapy (NST) in study participants. A false negative event will be defined as a case where the specific node (either the clipped node or the sentinel lymph node, depending on the analysis) does not show metastasis even though residual disease is identified in the other axillary nodes. The false negative rate will be computed as the number of false negative events divided by the total number of pathologically node-positive patients.

SECONDARY OUTCOMES:
Sentinel Lymph Node Identification Rate | Day 1 (Day of Surgery)
  The sentinel lymph node identification rate is the number of study participants with at least one sentinel lymph node divided by total number of study participants.
Clipped Lymph Node Identification Rate | Day 1 (Day of Surgery)
  The clipped lymph node identification rate is the number of study participants with at least one clipped lymph node removed divided by the total number of study participants with clipped lymph nodes.
Accuracy Rate of Imaging Studies | Up to 2 weeks
  The accuracy rate of imaging studies in determining response in the breast and axilla will be calculated as the sum of true responders on imaging and true non-responders on imaging divided by total number of study participants.
Pathologic Complete Response (pCR) | Up to 2 weeks
  The number of participants with pCR will be reported. The percentage of patients with pCR will be calculated as the number of patients with a pCR divided by the total number of study participants. PCR is defined as the lack of all signs of cancer in tissue samples removed during surgery.
Incidence of Treatment-Emergent Adverse Events | Up to 3 weeks
  Number of participants experiencing treatment-emergent adverse events (AEs). AEs will be assessed by and assigned severity and treatment attribution by the treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kesmodel, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No